CLINICAL TRIAL: NCT06894849
Title: Evaluation of a Text Message-Based Approach to Depression Screening Among Cancer Survivors
Brief Title: Text -Based Depression Screening Among Cancer Survivors
Acronym: OASIS1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Evan Graboyes, Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 00142039; FD006/CC001335/FN09 (Other Grant/Funding Number: Hollings Cancer Center)
Record Dates: First submitted 2025-02-06; First posted 2025-03-25 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Depression Secondary to Other Disease; Cancer Survivor
Keywords: Cancer Survivorship; Depression Screening; Text Message Screening; Mobile Health
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Text-Based Depression Screening (Experimental)
  Interventions: Behavioral: Text-based depression screening
- Usual Care (Active Comparator)
  Interventions: Behavioral: Usual care (UC)

INTERVENTIONS:
Behavioral: Text-based depression screening — Starting 1 week prior to the scheduled clinic appointment, patients will receive a text message invitation from HCC to complete depression screening. Participants will be asked to click to continue to the screening PHQ-2. For text message screening cadence, reminder texts will be sent daily for 3 days. Those who screen positive (PHQ-2 >/= 3) will complete the remainder of the items (i.e., PHQ-9).
  Arms: Text-Based Depression Screening
Behavioral: Usual care (UC) — Usual care (UC) will consist of in-person assessment of depression using a validated brief screening tool (e.g., PHQ-2) synchronous with a clinical encounter with the outpatient oncology team. Although the person completing the screening (e.g., nurse, medical assistant) and other workflow may vary slightly across settings, the 2-items are generally presented orally to the patient during routine intake for a clinical encounter and entered into the EHR. Patients who screen positive will be asked to complete the full PHQ-9.
  Arms: Usual Care

SUMMARY:
Depression is common among cancer survivors, but current screening methods are not always effective. To help improve depression screening for cancer survivors, this study will conduct a pilot randomized controlled trial (RCT) with 60 participants. The goal is to evaluate whether a text message-based approach to depression screening is feasible, acceptable, and potentially more effective than the current standard of care.

DETAILED DESCRIPTION:
This pilot randomized controlled trial aims to evaluate the feasibility, acceptability, and preliminary efficacy of a text message-based depression screening approach for cancer survivors. A total of 60 adult cancer survivors will be enrolled and randomly assigned to either the text message intervention or the usual care depression screening. The intervention involves sending text messages one week before scheduled oncology appointments, inviting participants to complete a depression screening using the PHQ-2, followed by the PHQ-9 for those who screen positive.

The study will assess the feasibility of implementing text message-based screenings, participant acceptability, and compare the efficacy of this method to traditional in-person depression screenings during clinical visits. The primary outcome is feasibility, measured by the proportion of participants completing the screening via text, while secondary outcomes will include acceptability (assessed through participant surveys) and preliminary efficacy (measured by screening completion rates and depression detection).

Eligible participants will be English-speaking cancer survivors aged 18 or older with an upcoming oncology appointment at the Hollings Cancer Center or associated clinics. The study aims to improve current depression screening methods and address challenges such as logistical and system-level barriers in screening cancer survivors for depression.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* diagnosis of cancer
* upcoming appointment in an HCC or HCN oncology clinic within 14 days
* English proficiency
* ownership of a cellphone with SMS text capability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Study Feasibility | 2 weeks after randomization
  >/= 1 response to a text message

SECONDARY OUTCOMES:
Acceptability | 2 weeks
  acceptability will be rated on a likert scale form 0-5 with higher scores representing greater acceptability
Depression screening | 2 weeks
  completion of PHQ-2 (Y/N)
PHQ-2 score | 2 weeks
  The PHQ-2 is a validated 2-item measure of depression screening that is widely used among patients with cancer. The PHQ-2 score ranges from 0 to 6. Higher scores indicate more severe depressive symptoms; a PHQ-2 score of ≥ 3 is considered a positive screening.
PHQ-9 score | 2 weeks
  Participants who screen positive for elevated depressive symptoms on the PHQ-2 (i.e, > 3) will complete the PHQ-9, a validated 9-item measure of depression. The PHQ-9 has high sensitivity and specificity for identifying individuals with depressive symptoms, particularly among cancer survivors. The PHQ-9 score ranges from 0 to 27; higher scores represent more severe depressive symptoms. A PHQ-9 score of ≥ 8 indicates clinically significant elevated depressive symptoms among patients with cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Evan Graboyes, MD, MPH, FACS, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided